CLINICAL TRIAL: NCT05168462
Title: Clinical Outcome and Cost-effectiveness of Reduced Noradrenaline by Using a Lower Blood Pressure Target in Patients With Cardiogenic Shock From Acute Myocardial Infarction
Acronym: NORSHOCK
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.P.S Henriques, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL79416.018.21
Record Dates: First submitted 2021-11-08; First posted 2021-12-23 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Cardiogenic Shock; Myocardial Infarction
Keywords: Noradrenaline; Blood pressure target; Cardiogenic shock; Myocardial infarction
MeSH Terms: conditions — Shock, Cardiogenic; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reduced noradrenaline (MAP ≥ 55 mmHg) (Experimental)
  Interventions: Drug: Reduced noradrenaline use
- Usual care (MAP ≥ 65 mmHg) (No Intervention)

INTERVENTIONS:
Drug: Reduced noradrenaline use — Reduced noradrenaline by using a lower MAP target
  Arms: Reduced noradrenaline (MAP ≥ 55 mmHg)

SUMMARY:
Rationale: Pump failure due to acute myocardial infarction (AMI) can lead to cardiogenic shock (CS): a state of low blood flow to end-organs with subsequent multi-organ failure that is associated with high mortality rated. The first line pharmacologic treatment strategy in CS is noradrenaline. This vasopressor drug is used to maintain adequate blood pressures. The assumption is that a mean arterial blood pressure (MAP) ≥ 65 mmHg will improve flow and thereby tissue perfusion of myocardium and other tissues (e.g. renal). However, there is no evidence that an increase in MAP, if achieved by noradrenaline, leads to greater end-organ blood flow and better outcomes.

Objective: With this study the investigators aim to investigate the (cost-)effectiveness of reduced noradrenaline in patients with CS by using a lower MAP target of ≥ 55 mmHg, compared to ≥ 65 mmHg. The investigators hypothesize that reduced use of noradrenaline will improve overall survival and decrease renal failure requiring renal replacement therapy.

Study design: Open label, randomized controlled multicenter trial

Study population: Adults patients with CS due to AMI

Intervention: Treatment strategy of reduced noradrenaline, by using a lower MAP target ( ≥ 55 mmHg).

Main study endpoint: composite of all-cause mortality and severe renal failure leading to renal replacement therapy within 30-days after randomization.

ELIGIBILITY:
Inclusion criteria:

1. Acute myocardial infarction, STEMI or NSTEMI
2. Early revascularization by PCI
3. Cardiogenic shock, characterized by:

I. a. Systolic blood pressure (SBP) ≤ 90 mmHg for > 30 minutes, OR b. Use of drugs to maintain SBP > 90 mmHg at randomization.

II. Clinical signs of impaired organ perfusion with at least one of the following criteria:

1. Altered mental status
2. Cold, clammy skin and extremities
3. Oliguria with urine output < 30ml/hour
4. Serum lactate > 2.0 mmol/L

III. Clinical signs of pulmonary congestion

Exclusion Criteria:

1. Resuscitation > 30 minutes
2. Mechanical cause of cardiogenic shock (e.g. papillary muscle rupture, ventricular septal rupture)
3. Onset of shock > 12 hours
4. Imminent need for mechanical circulatory support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 776 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Mortality and renal failure | 30-days
  Composite of all-cause mortality and severe renal failure leading to renal replacement therapy

SECONDARY OUTCOMES:
Blood pressure (systolic and diastolic) | The first 24 hours
  Blood pressure measured hourly during the first 24 hours of ICU/CCU admission
Heart rate | The first 24 hours
  Heart rate, measured hourly during the first 24 hours of ICU/CCU admission
Enzymatic infarct size, measured by hs-Troponin T | 0, 6, 12, 24, 36 and 72 hours
  Size of myocardial infarction, measured by hs-Troponin T
Enzymatic infarct size, measured by CK-MB | 0, 6, 12, 24, 36 and 72 hours
  Size of myocardial infarction, measured by CK-MB
Need for mechanical circulatory support | Recorded after ICU/CCU discharge, assessed up to 60 days
  Type of mechanical circulatory support device
Duration of mechanical ventilation | Recorded after ICU/CCU discharge, assessed up to 60 days
  Duration of mechanical ventilation, expressed in days
Need for vasopressors / inotropes | Recorded after ICU/CCU discharge, assessed up to 60 days
  The type of vasopressors / inotropes that were administrered
Ejection fraction, percent | 72 hours and 1 year
  As measured by echocardiography and/or MRI
Renal function | 1 year
  Renal function, measured by serum creatinin
Cost-effectiveness | 1-year
  Cost per patients alive without severe renal failure and costs per QALY (quality-adjusted life year)

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, location AMC, Amsterdam, Netherlands